CLINICAL TRIAL: NCT01022541
Title: Phase II Clinical Trial of Capecitabine and Oxaliplatin Plus Bevacizumab as Neoadjuvant Treatment for Patients With Previously Untreated Unresectable Liver-only Metastases From Colorectal Cancer
Brief Title: Capecitabine and Oxaliplatin Plus Bevacizumab as Neoadjuvant Treatment for Untreated Unresectable Liver-only Metastases From Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2676; NCT00450346 (obsolete NCT alias)
Record Dates: First submitted 2006-01-23; First posted 2009-12-01 (Estimated); Last update posted 2015-11-25 (Estimated); Status verified 2013-05

CONDITIONS: Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Capecitabine; Oxaliplatin; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- This is a single arm study (Other): This is a single arm study
  Interventions: Drug: Capecitabine; Drug: Oxaliplatin; Drug: Bevacizumab; Procedure: Liver metastasectomy

INTERVENTIONS:
Drug: Capecitabine — Capecitabine 1700mg/m2/day in two divided doses to be administered orally for 14 days followed by 7 days rest. For 4 courses initially.
  (For patients aged 75+ 1300mg/m2/day in two divided doses or 650mg/m2 twice daily)
  Courses as per detailed description above.
  Other Names: Xeloda
Drug: Oxaliplatin — Oxaliplatin 130mg/m2 diluted in 5% dextrose will be given as an i.v. infusion over 2 hours. This will be administered on day 1 after bevacizumab. For 4 courses.
  (Patients aged 75+ should receive oxaliplatin at a reduced dose i.e. 100mg/m2)
  Courses as per detailed description above.
  Other Names: Eloxatin
Drug: Bevacizumab — Bevacizumab at a dose of 7.5 mg/kg, diluted in normal saline, will be administered as an iv infusion over 30 to 90 minutes before the administration of oxaliplatin on day 1 of every cycle.
  The first infusion should be administered over 90 minutes. If well tolerated, the second infusion can be administered over 60 minutes. Provided that this is tolerated subsequent infusions can be administered over 30 minutes. If a patient experiences an infusion related adverse event with the 60 minute infusion, all subsequent infusions will be administered over 90 minutes. If a patient experiences an infusion related reaction with the 30 minute infusion, all subsequent infusions will be administered over 60 minutes
  Courses as per detailed description above.
  Other Names: Avastin
Procedure: Liver metastasectomy — Patients with liver metastases which have become resectable and in whom surgery is still deemed appropriate should proceed to surgery after a 6 week interval from the last administration of capecitabine chemotherapy (at least 8 weeks from last administration of bevacizumab).

SUMMARY:
To evaluate the overall response rate of patients with previously untreated unresectable liver-only metastases from colorectal cancer treated with neoadjuvant capecitabine and oxaliplatin plus bevacizumab.

DETAILED DESCRIPTION:
No previous treatment.

The 21 day cycle of treatment will be given for four courses before being reassessed by MRI/CT for resectability of their liver metastases.

Those patients with stable disease or partial response, but are not yet resectable will continue for a further four courses of treatment before reassessment.

Patients whose liver metastases have become resectable will proceed to surgery after a 6 week break from the last administration of Capecitabine (8 weeks from the last administration of Bevacizumab).

A further four courses of treatment will be administered post-operatively to commence at least 8 weeks after surgery and when the patient is well recovered and healed.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven diagnosis of colorectal adenocarcinoma
* Metastatic disease present in the liver only.
* Absence of extrahepatic metastases excluded by CT chest, abdomen and pelvis. Indeterminate CT findings may require verification by FDG-PET scanning.
* Liver-only metastases determined to be unresectable at presentation on a pre-treatment liver MRI with an appropriate liver specific contrast (eg. TESLA) by a specialist multidisciplinary team (consisting of medical oncologist, hepatic surgeon and radiologist). Guidelines for determining unresectability include:
* presence of >4 metastases;
* size >5cm;
* location and distribution of metastatic disease within the liver unsuitable for resection with clear margins (eg. Involvement of both lobes of liver; invasion of intrahepatic vascular structures);
* extent of liver involvement precluding resection with adequate post-resection residual liver parenchyma volume for viable liver function in the immediate post-operative period;
* inability to retain adequate vascular in flow and out flow to maintain viable liver function.
* No previous treatment for metastatic colorectal cancer, including chemotherapy, targeted or experimental therapies (e.g. anti-VEGF or anti-EGFR), radiotherapy to the liver, or surgery or radiofrequency ablation to liver metastases.
* Feasibility of surgery with curative intent:
* If the primary colorectal tumour is in situ, the primary tumour must also be resectable with curative intent
* Patients presenting with liver metastases only relapse after initially curative resection of their primary colorectal cancer followed by treatment with adjuvant chemotherapy may not be entered into the study if the relapse has occurred within 12 months of completion of adjuvant treatment
* Adequate medical fitness to undergo neoadjuvant treatment and surgery with curative intent (hepatectomy +/- resection of primary tumour, if required)
* Absence of pre-existing liver dysfunction of Childs Pugh Grade B or greater. Patients who are suspected of having pre-existing liver dysfunction due to clinical, biochemical or radiological findings, should have significant liver disease excluded by a liver biopsy prior to study entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2006-06; Primary Completion 2010-12 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Overall response rates | 12 months

SECONDARY OUTCOMES:
Complete resection (R0) rate | 12 months
Safety and feasibility of adding bevacizumab to neoadjuvant capecitabine and oxaliplatin in patients undergoing liver metastasectomy | 12 months
Other parameters of efficacy (response and survival) in patients with unresectable liver-only metastases treated with this neoadjuvant combination | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: David Cunningham, Principal Investigator — Royal Marsden NHS Foundation Trust
Locations (1):
- David Cunningham, Sutton, Surrey, United Kingdom

REFERENCES:
- [Derived] Wong R, Cunningham D, Barbachano Y, Saffery C, Valle J, Hickish T, Mudan S, Brown G, Khan A, Wotherspoon A, Strimpakos AS, Thomas J, Compton S, Chua YJ, Chau I. A multicentre study of capecitabine, oxaliplatin plus bevacizumab as perioperative treatment of patients with poor-risk colorectal liver-only metastases not selected for upfront resection. Ann Oncol. 2011 Sep;22(9):2042-2048. doi: 10.1093/annonc/mdq714. Epub 2011 Feb 1. PMID 21285134